CLINICAL TRIAL: NCT01843855
Title: The Contribution of Incretin Hormones to the Amelioration of Glucose Metabolism After Roux-en-Y Gastric Bypass
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Adrian Vella (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor-Investigator, Adrian Vella, Consultant, Endocrinology, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 11-000161; R01DK082396 (NIH); UL1RR024150 (NIH)
Record Dates: First submitted 2013-04-26; First posted 2013-05-01 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-12

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Gastric Bypass; bariatric surgery; glucose metabolism
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exendin 9,39 (Experimental): Subjects randomized to this arm will receive an infusion of exendin 9,39 of 300mmol/kg/min for 360 minutes.
  Interventions: Drug: Exendin 9,39
- Placebo (Placebo Comparator): Subjects randomized to this arm will receive a saline infusion for 360 minutes.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Exendin 9,39 — Exendin 9,39 is a competitive antagonist of endogenous GLP-1.
  Arms: Exendin 9,39
Drug: Placebo — A saline infusion will be given to match the study drug infusion.
  Arms: Placebo

SUMMARY:
The study is being undertaken to understand how a gastric bypass can affect a subject's diabetes even prior to their losing significant amounts of weight. The hypothesis of this study is that increased glucagon-like peptide-1 (GLP-1) secretion explains the amelioration in insulin secretion after Roux-en-Y Gastric Bypass (RYGB) surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with type 2 diabetes mellitus or impaired fasting glucose concentration of > 110 mg/dL
* Subjects registered to receive a Roux-en-Y Gastric Bypass (RYGB).

Exclusion Criteria:

* Subjects taking thiazolidinediones
* Subjects with active systemic illness
* Subjects with active microvascular or macrovascular complications of their diabetes
* For female subject: positive pregnancy test at the time of enrollment in study

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-06; Primary Completion 2013-07 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Change in Total Disposition Index from Study 1 (pre-RYGB) to Study 2 (post-RYGB) | baseline, 4 weeks post-operative intervention
  The total disposition index equals the product of insulin secretion and insulin sensitivity.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Vella, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States